CLINICAL TRIAL: NCT01800578
Title: Relationships Between Bispectral Index (BIS), Implicit Memory Dream Recall and MAC in Blended Anaesthesia
Brief Title: Awareness During Blended Anaesthesia
Status: Completed | Type: Observational
Sponsor: Germano De Cosmo (Other)
Responsible Party: Sponsor-Investigator, Germano De Cosmo, PhD, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Other Study IDs: A1044/2001
Record Dates: First submitted 2012-11-12; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Consciousness, Level Depressed; Intraoperative Awareness
Keywords: Cerebral State Index Monitor
MeSH Terms: conditions — Consciousness Disorders; Intraoperative Awareness | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bispectral Index Group
  Interventions: Device: monitor for depth of hypnosis

INTERVENTIONS:
Device: monitor for depth of hypnosis — evaluation of depth of hypnosis
  --------------------------------------------------------------------------------

SUMMARY:
the aim of this study was to estimate the relations between Bispectral Index values and explicit or implicit memory or dreams during two different minimal alveolar concentration (MAC) of sevoflurane in patients undergoing blended anaesthesia for major abdominal surgery and ,in this way, estimate the possibility to reduce, in presence of a deep analgesia, like epidural analgesia, the requirement of halogenated volatile anesthetics.

DETAILED DESCRIPTION:
The decreased responsiveness to stimulation defines depth of anaesthesia which is a balance between effects of anaesthetic drugs and surgical stimulations.

Awareness is a rare occurrence with an incidence of 0,1-0,2 % , defined as postoperative recall of events occurring during general anaesthesia.

Different stages of awareness should be defined: conscious awareness with explicit recalls with pain; conscious awareness with explicit recalls without pain; conscious awareness without explicit recall and possible implicit recall; subconscious awareness without explicit recall and possible implicit recall; no awareness .

This memory can be traumatic and may result in developing a chronic posttraumatic stress disorder (PTSD) in more than half of subjects .

Some cases of awareness are caused by inadequate anesthesia and are potentially avoidable through the assessment of depth of hypnosis by an intraoperative monitoring , especially when muscle relaxants are used.

The Bispectral Index ( BIS ), one of the devices designed to monitor brain activity, through a proprietary algorithm , elaborates EEG and provides an index of hypnotic level.

Thus, several variables, derived from EEG time and frequency domain, are combined into a single index indicating the patient's level of consciousness.

A range between 40 and 60, during surgery, permits both to prevent awareness and to reduce the dose of anesthetic agent administered .

In this study, during major abdominal surgery, an epidural analgesia was performed to suppress afferent noxious stimuli and combined with a general anaesthesia based on halogenates.

Thereby the aim of this study was to estimate the relations between Bispectral Index values and explicit or implicit memory or dreams during two different minimal alveolar concentration (MAC) of sevoflurane in patients undergoing blended anaesthesia for major abdominal surgery and ,in this way, estimate the possibility to reduce, in presence of a deep analgesia, like epidural analgesia, the requirement of halogenated volatile anesthetics.

ELIGIBILITY:
Inclusion Criteria:

native Italian speakers American society of anaesthesiologist physical status I-II -

Exclusion Criteria:refusal of placement of epidural catheter neurological or psychiatric diseases hearing impairment use of drugs know to affect central nervous system coagulopathy heart conditions infections allergy to local anaesthetics liver or renal disease

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
correlation between BIS and free association test score | every 15 min during anaesthesia and 24 h after emergency from anaesthesia

SECONDARY OUTCOMES:
MAC of sevoflurane necessary to avoid awareness | 24 h after emergency from anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: De Cosmo Germano, PhD, Principal Investigator — Catholic University
Locations (1):
- Catholic University of Sacred Heart, Rome, Rm, Italy

REFERENCES:
- [Background] Wong CS. What's the matter of depth of anesthesia? Acta Anaesthesiol Sin. 2001 Mar;39(1):1-2. No abstract available. PMID 11407288
- [Background] Sandin RH, Enlund G, Samuelsson P, Lennmarken C. Awareness during anaesthesia: a prospective case study. Lancet. 2000 Feb 26;355(9205):707-11. doi: 10.1016/S0140-6736(99)11010-9. PMID 10703802
- [Background] Schwender D, Klasing S, Daunderer M, Madler C, Poppel E, Peter K. [Awareness during general anesthesia. Definition, incidence, clinical relevance, causes, avoidance and medicolegal aspects]. Anaesthesist. 1995 Nov;44(11):743-54. doi: 10.1007/s001010050209. German. PMID 8678265
- [Background] Osterman JE, Hopper J, Heran WJ, Keane TM, van der Kolk BA. Awareness under anesthesia and the development of posttraumatic stress disorder. Gen Hosp Psychiatry. 2001 Jul-Aug;23(4):198-204. doi: 10.1016/s0163-8343(01)00142-6. PMID 11543846
- [Background] Baars BJ. The brain basis of a "consciousness monitor": scientific and medical significance. Conscious Cogn. 2001 Jun;10(2):159-64; discussion 246-58. doi: 10.1006/ccog.2001.0510. PMID 11414712
- [Background] Ghoneim MM. Incidence of and risk factors for awareness during anaesthesia. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):327-43. doi: 10.1016/j.bpa.2007.05.002. PMID 17900012
- [Background] Ekman A, Lindholm ML, Lennmarken C, Sandin R. Reduction in the incidence of awareness using BIS monitoring. Acta Anaesthesiol Scand. 2004 Jan;48(1):20-6. doi: 10.1111/j.1399-6576.2004.00260.x. PMID 14674969
- [Background] Aceto P, Valente A, Gorgoglione M, Adducci E, De Cosmo G. Relationship between awareness and middle latency auditory evoked responses during surgical anaesthesia. Br J Anaesth. 2003 May;90(5):630-5. doi: 10.1093/bja/aeg113. PMID 12697591